CLINICAL TRIAL: NCT06352606
Title: Comparison Between Spinal and General Anesthesia in Neonates Undergoing Herniorrhaphy: A Randomized Controlled Trial
Brief Title: Spinal and General Anesthesia in Neonates Undergoing Herniorrhaphy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 36264PR558/2/24
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Spinal Anesthesia; General Anesthesia; Neonates; Inguinal Herniorrhaphy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Anesthesia (Experimental): Oxygen supply will be done via nasal prong (2 L/min) when necessary. The local anesthetic used will be bupivacaine 0.6 mg/kg.
  Interventions: Diagnostic Test: Spinal anesthesia
- General Anesthesia (Active Comparator): Patients will receive sevoflurane for induction and maintenance in an air/oxygen mixture along. Endotracheal tube will be inserted. No opioids or nitrous oxide was used intraoperatively.
  Interventions: Diagnostic Test: General anesthesia

INTERVENTIONS:
Diagnostic Test: Spinal anesthesia — Oxygen supply will be done via nasal prong (2 L/min) when necessary. The local anesthetic used will be bupivacaine 0.6 mg/kg.
  Arms: Spinal Anesthesia
Diagnostic Test: General anesthesia — Patients will receive sevoflurane for induction and maintenance in an air/oxygen mixture along. Endotracheal tube will be inserted. No opioids or nitrous oxide was used intraoperatively.
  Arms: General Anesthesia

SUMMARY:
The aim of this study is to compare spinal and general anesthesia in neonates undergoing herniorrhaphy.

DETAILED DESCRIPTION:
Spinal anesthesia (SA) is a fast, simple and cost-effective method that has been used for the performance of inguinal hernias since the beginning of the 20th century in adults.

One large observational study documented a low risk of post operative events with spinal anesthesia for inguinal hernia repair in infants . In addition, a randomized trial comparing reginal and general anesthesia in this population have not shown any significant differences in outcome. Spinal anesthesia reduces postoperative oxygen desaturation and respiratory morbidity when compared to general anesthesia (GA) in infants who underwent inguinal herniorrhaphy

ELIGIBILITY:
Inclusion Criteria:

* Neonates either full term or preterm.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II
* Undergoing unilateral or bilateral inguinal herniorrhaphy.

Exclusion Criteria:

* Obstructed hernia.
* Neonates with significant chronic lung disease (e.g., disease associated with hypoxemia in room air or chronic hypercapnia).
* Symptomatic congenital heart disease (e.g., cyanosis or congestive heart failure).
* Symptomatic central nervous system disease (e.g., seizures).

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Immediately postoperatively at post-anesthesia care unit
  Heart rate will be recorded at post-anesthesia care unit.

SECONDARY OUTCOMES:
Heart rate | Till two hours postoperatively
  Heart rate will be recorded at baseline, every 10 min intraoperatively and every 30 min in post-anesthesia care unit.
Mean arterial blood pressure | Till two hours postoperatively
  Mean arterial blood pressure will be recorded at baseline, every 10 min intraoperatively and every 30 min in post-anesthesia care unit.
Incidence of bradycardia | 24 hours postoperative
  Incidence of bradycardia will be measured, defined by decrease in basal heart rate by 20% and will be treated by I.V. atropine 0.02 mg/kg.
Incidence of hypotension | 24 hours postoperative
  Hypotension will be assessed
Incidence of postoperative apnea | 24 hour postoperatively
  Apnea is defined as a pause in breathing for more than 15 s or more than 10 s if associated with oxygen saturation less than 80% or bradycardia (20% decrease in heart rate). Early apnea is defined as a priori as an apnea occurring within the first 30min postoperatively in the PACU, and late apnea is defined as an observed apnea occurring between 30 min and 12 hour postoperatively.
The duration of surgery | Till the end of surgery
  The duration of surgery will be assessed from the start of surgery till the end of surgery.
Need for postoperative O2 supplementation | Till two hours postoperatively
  Oxygen saturation will be recorded at baseline, every 10min intraoperatively and every 30 min in post-anesthesia care unit (PACU).
Hospital stays | 28 days postoperative
  Hospital stays will be assessed from admission till discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author